CLINICAL TRIAL: NCT04730817
Title: Virtual Reality Motor-cognitive Training for Older People With Cognitive Frailty: The Implementation of the Prototype
Brief Title: VR Motor-cognitive Training for Older People With Cognitive Frailty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Pok Oi Hospital (Other)
Responsible Party: Principal Investigator, Dr Rick Kwan, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K-ZB1H
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Cognitive Frailty; Physical Function
Keywords: Cognitive Frailty; Motor-Cognitive Training; Virtual Reality; Gamification

STUDY DESIGN:
Intervention Model Description: A total of 400 subjects with cognitive frailty will be assigned into 2 groups. Half the participants will be assigned to the intervention group in which they will undertake VR simultaneous motor-cognitive training and others will be assigned to the control group in the form of passive (wait list) control, i.e., they will not be given any kind of treatment.
  The following dosage will be employed onto the intervention group using the VR simultaneous motor-cognitive training that we proposed. I.e.,
  Course: eight weeks Session duration: 30 minutes Frequency: twice per week
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors at both pre- and post-observations will be blinded to the group label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This arm will undertake VR simultaneous motor-cognitive training in 30 minutes session, twice a week for 8 weeks.
  Interventions: Device: Virtual Reality Motor-Cognitive Training System
- Control group (No Intervention): This arm will not be given any kind of treatment and will act as a passive control group.

INTERVENTIONS:
Device: Virtual Reality Motor-Cognitive Training System — Immersive VR training system tailor-made for the daily living experiences in the Hong Kong context to provide interactive experiences for older people in Hong Kong. The VR training system is designed as a game with 16 progressive levels (anticipating intervention group participants to complete 2 levels per week for 8 weeks) which aim to train their motor and cognitive functions.
  Arms: Intervention group

SUMMARY:
Cognitive frailty is a clinical syndrome in which cognitive impairment (e.g., poor memory, visuospatial function) and physical frailty (e.g., slowness, poor muscle strength, physical inactivity) co-exist. It is prevalent in community-dwelling older people. The progressive decline of cognitive and physical functions restricts older people from participating in activities (e.g., social get-togethers). Reduced participation further jeopardizes their life-space mobility (e.g., ability to travel to areas far away from home). Therefore, those with cognitive frailty are at risk of developing dementia and becoming dependent.

Simultaneous motor-cognitive training is more effective at promoting optimal functioning in older people than motor or cognitive training alone. Gaming is effective at promoting the motivation to participate. The contents of games in the market are unrelated to the context or daily living of the elderly. Currently, available training is non-simultaneous. This makes the training less transferable to the daily life of the elderly and reduces its effects.

Virtual reality (VR) technology can provide a virtual space that mimics the real environment. This allows clients to participate in daily activities in a virtual space. Older people can be trained to improve their cognitive and physical skills in a painless, fun way. However, the effect and feasibility of employing simultaneous motor-cognitive training launching on a VR platform mimicking the daily living environment in older people with cognitive frailty is poorly known.

Following the findings from the previous proof-of-concept test (registration number: NCT04467216), we proceed to implement the study to 400 participants from six different elderly centres between the period of March 2021 and December 2022.

DETAILED DESCRIPTION:
In the intervention, VR will be employed to simulate a daily living environment familiar to older people. Participants will wear a commercially available head-mounted VR system with hand-held controllers to experience the participation of daily activities in a virtual environment. Simultaneous physical and cognitive training will be embedded in the training system to promote optimal function. Participants will attend physical training in a sitting position through cycling on an ergometer and moving the hand-held controllers. Motion sensors built into the VR system and ergometer will track these movements to control everyday tasks in the virtual environment (e.g., moving around the city). Simultaneously, participants will undergo cognitive training by participating in various tasks demanding cognitive functions, such as visual-spatial (e.g., wayfinding) and problem-solving (e.g., wallet loss) functions. Gamification will be employed to promote the motivation to participate. All training activities will be gamified by blending in fun elements, such as difficulty-levelling, competition, and e-tokens. Co-participation is allowed to promote interpersonal interactions. The prototype enables real-time co-viewing among participants. Other elderly centre members and the activity facilitators can share the view of the participants in the game on either a large-screen monitor or a tablet computer, allowing them to simultaneously discuss and share about their gaming experiences.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years,
* Self-reported or informant-reported cognitive complaints
* Objective cognitive impairment, as defined by a Clinical Dementia Rating of 0.5 and a Montreal Cognitive Assessment (MoCA) score of <25
* Preservation of one's independence, as defined by the Lawton's Instrumental Activity of Daily Living score of >14
* No diagnosed dementia, as observed in the medical record
* Physical frailty from being pre-frail to frail, as defined by a Fried Frailty Index (FFI) score of 1-5.

Exclusion Criteria:

* Participants who have impaired mobility, as defined by Modified Functional Ambulatory Classification (MFAC) < Category 7 (i.e., Outdoor walker),
* or probable dementia, i.e., MoCA < 17 or clinical dementia rating ≥ 1.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Global cognitive function | Change is being assessed at "baseline" (T0) and "immediately after the completion" (T1), being 8 weeks apart
  Score on the Montreal Cognitive Assessment Hong Kong Version (HK-MoCA), ranging from 0 to 30.
Frailty | Change is being assessed at "baseline" (T0) and "immediately after the completion" (T1), being 8 weeks apart
  Score on the Fried Frailty Phenotype, ranging from 0 to 5

SECONDARY OUTCOMES:
Inhibition of cognitive interference | Change is being assessed at "baseline" (T0) and "immediately after the completion" (T1), being 8 weeks apart
  Stroop Color-Word Test (SCWT) Global Index score, calculated by I=CW-((W+C)/2)
Executive function | Change is being assessed at "baseline" (T0) and "immediately after the completion" (T1), being 8 weeks apart
  Time taken to complete the trail making test (TMA & TMB), ranges from 0 to 300 seconds (when maximum time is reached)
Verbal and visuo-spatial short-term memory | Change is being assessed at "baseline" (T0) and "immediately after the completion" (T1), being 8 weeks apart
  Score on the Digit Span Test, ranges from 0 to 9
Walking speed | Change is being assessed at "baseline" (T0) and "immediately after the completion" (T1), being 8 weeks apart
  Timed up and go test (seconds)
Hand grip strength | Change is being assessed at "baseline" (T0) and "immediately after the completion" (T1), being 8 weeks apart
  Hand grip strength by dynamometer (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Rick Kwan, Dr, Principal Investigator — The Hong Kong Polytechnic University
Locations (6):
- Hong Kong (6):
  - Pok Oi Hospital Chan Shi Sau Memorial Social Service Centre, Hong Kong
  - Pok Oi Hospital Mei Foo Lai Wan Kaifong Association Mr. and Mrs. Leung Chi Chim Elderly Health Support and Learning Centre, Lai Chi Kok
  - Pok Oi Hospital Mr. Kwok Hing Kwan Neighbourhood Elderly Centre, Lai Chi Kok
  - Pok Oi Hospital Chan Ping Memorial Neighbourhood Elderly Centre, Tin Shui Wai
  - Pok Oi Hospital Wong Muk Fung Memorial Elderly Health Support and Learning Centre, Tuenmen
  - Pok Oi Hospital Mrs. Wong Tung Yuen District Elderly Community Centre, Yuen Long

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruan Q, Yu Z, Chen M, Bao Z, Li J, He W. Cognitive frailty, a novel target for the prevention of elderly dependency. Ageing Res Rev. 2015 Mar;20:1-10. doi: 10.1016/j.arr.2014.12.004. Epub 2014 Dec 30. PMID 25555677
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Wong A, Xiong YY, Kwan PW, Chan AY, Lam WW, Wang K, Chu WC, Nyenhuis DL, Nasreddine Z, Wong LK, Mok VC. The validity, reliability and clinical utility of the Hong Kong Montreal Cognitive Assessment (HK-MoCA) in patients with cerebral small vessel disease. Dement Geriatr Cogn Disord. 2009;28(1):81-7. doi: 10.1159/000232589. Epub 2009 Aug 11. PMID 19672065
- [Background] Yeung PY, Wong LL, Chan CC, Leung JL, Yung CY. A validation study of the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) in Chinese older adults in Hong Kong. Hong Kong Med J. 2014 Dec;20(6):504-10. doi: 10.12809/hkmj144219. Epub 2014 Aug 15. PMID 25125421
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Viosca E, Martinez JL, Almagro PL, Gracia A, Gonzalez C. Proposal and validation of a new functional ambulation classification scale for clinical use. Arch Phys Med Rehabil. 2005 Jun;86(6):1234-8. doi: 10.1016/j.apmr.2004.11.016. PMID 15954065
- [Background] Kelaiditi E, Cesari M, Canevelli M, van Kan GA, Ousset PJ, Gillette-Guyonnet S, Ritz P, Duveau F, Soto ME, Provencher V, Nourhashemi F, Salva A, Robert P, Andrieu S, Rolland Y, Touchon J, Fitten JL, Vellas B; IANA/IAGG. Cognitive frailty: rational and definition from an (I.A.N.A./I.A.G.G.) international consensus group. J Nutr Health Aging. 2013 Sep;17(9):726-34. doi: 10.1007/s12603-013-0367-2. PMID 24154642
- [Background] Desjardins-Crepeau L, Berryman N, Fraser SA, Vu TT, Kergoat MJ, Li KZ, Bosquet L, Bherer L. Effects of combined physical and cognitive training on fitness and neuropsychological outcomes in healthy older adults. Clin Interv Aging. 2016 Sep 19;11:1287-1299. doi: 10.2147/cia.s115711. eCollection 2016. PMID 27698558
- [Background] Lauenroth A, Ioannidis AE, Teichmann B. Influence of combined physical and cognitive training on cognition: a systematic review. BMC Geriatr. 2016 Jul 18;16:141. doi: 10.1186/s12877-016-0315-1. PMID 27431673
- [Background] Tait JL, Duckham RL, Milte CM, Main LC, Daly RM. Influence of Sequential vs. Simultaneous Dual-Task Exercise Training on Cognitive Function in Older Adults. Front Aging Neurosci. 2017 Nov 7;9:368. doi: 10.3389/fnagi.2017.00368. eCollection 2017. PMID 29163146
- [Background] de Vries AW, Faber G, Jonkers I, Van Dieen JH, Verschueren SMP. Virtual reality balance training for elderly: Similar skiing games elicit different challenges in balance training. Gait Posture. 2018 Jan;59:111-116. doi: 10.1016/j.gaitpost.2017.10.006. Epub 2017 Oct 5. PMID 29028622
- [Background] Scarpina F, Tagini S. The Stroop Color and Word Test. Front Psychol. 2017 Apr 12;8:557. doi: 10.3389/fpsyg.2017.00557. eCollection 2017. PMID 28446889
- [Background] Monaco M, Costa A, Caltagirone C, Carlesimo GA. Forward and backward span for verbal and visuo-spatial data: standardization and normative data from an Italian adult population. Neurol Sci. 2013 May;34(5):749-54. doi: 10.1007/s10072-012-1130-x. Epub 2012 Jun 12. PMID 22689311
- [Background] Wei M, Shi J, Li T, Ni J, Zhang X, Li Y, Kang S, Ma F, Xie H, Qin B, Fan D, Zhang L, Wang Y, Tian J. Diagnostic Accuracy of the Chinese Version of the Trail-Making Test for Screening Cognitive Impairment. J Am Geriatr Soc. 2018 Jan;66(1):92-99. doi: 10.1111/jgs.15135. Epub 2017 Nov 14. PMID 29135021
- [Background] Freitas S, Simoes MR, Alves L, Santana I. Montreal cognitive assessment: validation study for mild cognitive impairment and Alzheimer disease. Alzheimer Dis Assoc Disord. 2013 Jan-Mar;27(1):37-43. doi: 10.1097/WAD.0b013e3182420bfe. PMID 22193353
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Tong AYC, Man DWK. The Validation of the Hong Kong Chinese Version of the Lawton Instrumental Activities of Daily Living Scale for Institutionalized Elderly Persons. OTJR: Occupation, Participation and Health. 2002; 22(4): 132-142.
- [Background] Chau MWR, Chan SP, Wong YW, Lau MYP. Reliability and validity of the Modified Functional Ambulation Classification in patients with hip fracture. Hong Kong Physiotherapy Journal. 2013; 31(1): 41-44.
- [Derived] Kwan RYC, Liu J, Sin OSK, Fong KNK, Qin J, Wong JCY, Lai C. Effects of Virtual Reality Motor-Cognitive Training for Older People With Cognitive Frailty: Multicentered Randomized Controlled Trial. J Med Internet Res. 2024 Sep 11;26:e57809. doi: 10.2196/57809. PMID 39259959